CLINICAL TRIAL: NCT03880162
Title: Metabolic Effects of a Low Carbohydrate Versus Energy-matched Standard Diet in Morbidly Obese Individuals With Prediabetes
Brief Title: Metabolic Effects of a Low Carbohydrate Versus a Standard Diet in Morbidly Obese With Prediabetes
Acronym: CaPrO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CaPrO
Record Dates: First submitted 2019-03-07; First posted 2019-03-19 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: PreDiabetes; Obesity, Morbid; Bariatric Surgery Candidate
Keywords: Prediabetes; Bariatric Surgery; Low-carb diet
MeSH Terms: conditions — Prediabetic State; Obesity, Morbid | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Intervention Model Description: Single-centre, randomized parallel study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study intervention (Experimental): Participants will follow an energy deficient (30% deficit) low carbohydrate diet (10% of carbohydrates) for minimum two weeks.
  Interventions: Other: Low carbohydrate diet
- Control intervention (Active Comparator): Participants will follow an energy deficient (30% deficit) standard diet (50% of carbohydrates) for minimum two weeks.
  Interventions: Other: Energy-matched standard diet

INTERVENTIONS:
Other: Low carbohydrate diet — A energy deficient (30% deficit) low carbohydrate diet (10% of carbohydrates)
  Arms: Study intervention
Other: Energy-matched standard diet — Energy-matched (30% deficit) standard diet (50% of carbohydrates)
  Arms: Control intervention

SUMMARY:
To investigate the metabolic effects of a low carbohydrate versus energy-matched standard diet in morbidly obese individuals with prediabetes awaiting bariatric surgery.

DETAILED DESCRIPTION:
The metabolic benefits of calorie restriction in obese people with or without impaired glycaemia are well-established. The impact of diet composition, however, remains poorly understood. Hepatic lipid content strongly correlates with hepatic insulin resistance, which is a key feature of the pre-diabetic state. The investigators hypothesize that a low carbohydrate diet compared to an energy-matched standard diet in morbidly obese patients with prediabetes scheduled for bariatric surgery results in greater reduction in liver fat.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects aged 18 years or older
* BMI >35 kg/m2 awaiting bariatric surgery
* Pre-diabetes according to American Diabetes Association criteria (HbA1c 5.7%-6.4%)
* Capacity to give informed consent and adhere to study procedures

Exclusion Criteria:

* Excess alcohol consumption (> 3 units/day for men, > 2 units/day for women)
* Moderate to severe kidney disease
* Nephrolithiasis
* Pregnancy/breastfeeding
* Current participation in another clinical trial
* Claustrophobia
* MRI-contraindications (pacemaker/defibrillator, neurostimulator, drug pump, cochlear implant, heart valve/vascular clips, shunt valve)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in intrahepatic triglyceride content | 2 weeks
  The intrahepatic triglyceride content will be evaluated by magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Change from baseline in body weight | 2 weeks
  The body weight will be measured using a pre-defined person scale
Change from baseline in liver size | 2 weeks
  The liver size will be evaluated by magnetic resonance imaging
Change from baseline in visceral adipose tissue | 2 weeks
  The adipose tissue content will be evaluated by magnetic resonance imaging
Change from baseline in whole body fat mass | 2 weeks
  Fat mass will be evaluated by bioimpedance
Change from baseline in insulin secretion | 2 weeks
  The insulin secretion will be evaluated during an oral glucose tolerance test using the oral minimal model
Change from baseline in insulin sensitivity | 2 weeks
  The insulin sensitivity will be evaluated during an oral glucose tolerance test using the oral minimal model

OTHER OUTCOMES:
Change from baseline in plasma metabolome | 2 weeks
  Fasting serum sampling
Change from baseline in plasma transcriptome | 2 weeks
  Fasting serum sampling
Change from baseline in Fibroblast Growth Factor 21 | 2 weeks
  Plasma level
Change from baseline in adipose tissue inflammation | 2 weeks
  Adipose tissue histology
Change from baseline in gut microbiota composition | 2 weeks
  Distribution of the predominant bacterial phylotypes will be assessed after 16S rRNA amplicon sequencing and subsequent taxonomic classification
Change from baseline levels of secondary bile acids | 2 weeks
  Faecal sampling
Change in frequency of immune cells (T-, B-, NK-cells, monocytes, neutrophils) | 2 weeks
  Frequency of immune cells will be analysed using flowcytometry
Change in immunometabolism of T-cells | 2 weeks
  Immunometabolism will be assessed by quantifying rates of oxygen consumption and glycolysis using metabolic flux analysis
Occurrence of surgical complication | Day of surgery until 2 weeks post-surgery
  Occurrence of the following: anastomotic leak, infection, bleeding, deep venous thrombosis (based on medical records)
Length of hospital stay | Day of surgery until 2 weeks post-surgery
  Based on medical records

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD PhD, Principal Investigator — Inselspital, Bern University Hospital, University of Bern
Locations (1):
- Division of Endocrinology, Diabetes and Clinical Nutrition, Bern University Hospital, Bern, Switzerland